CLINICAL TRIAL: NCT00634868
Title: Treatment of Wounds Utilizing Light
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow patients recruitment
Sponsor: QRay Ltd. (Industry)
Responsible Party: Qray Ltd, Qray
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: or003121107
Record Dates: First submitted 2008-02-07; First posted 2008-03-13 (Estimated); Last update posted 2011-06-10 (Estimated); Status verified 2011-06

CONDITIONS: Diabetic Ulcer
Keywords: ulcer wound diabetes

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Sham Comparator): The device is emitting a sham light
  Interventions: Device: Qray light therapy device-Sham
- 2 (Experimental): The device is emitting curative light
  Interventions: Other: Qray light therapy device

INTERVENTIONS:
Other: Qray light therapy device — The light is filtered from harmful UV and InfraRed light and only light at wavelight of 405nm until 1000nm is delivered.
  Arms: 2
Device: Qray light therapy device-Sham — non curative light- the device emits the same broad light, but with very low intensity
  Arms: 1

SUMMARY:
The Qray device is emitting broad light energy that is intended for diabetic ulcer healing. The study is double blinded.

ELIGIBILITY:
Inclusion Criteria:

* Patient has 8 weeks venus leg ulcer.
* The ulcer was not better on prior treatment of various medical clinics.
* The patient has diabetic ulcer grade 1 or 2

Exclusion Criteria:

* Patient has severe infection.
* Patient is taking antibiotic
* Patient has ankle brachial index less than 0.7
* Patient is schedule to undergone revascularization surgery 10 weeks before the study
* Patient has photosensitive disease
* Patient has cancer
* Creatinine level is more than 2 mg%
* Patient is taking immunosuppressive medication.
* Pregnant women
* Dialysis patient
* Anaemic patients(less than 9 gr)
* Patient has Albumin level less than 3 mg%

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2008-08; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
The wound healing process | 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Soroka Medical Center, Beersheba, Israel